CLINICAL TRIAL: NCT02374723
Title: Evaluation of Biosynthetic Constructs as Replacement for Donor Corneas as Graft Material for Corneal Transplantation
Brief Title: Evaluation of Biosynthetic Constructs to Replace Donor Corneas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was withdrawn to be replaced with a multi-site Phase I trial.
Sponsor: Region Östergötland (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Per.Fagerholm, professor,MD,PhD, Region Östergötland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNr52120125706
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Corneal Disease
Keywords: improve; vision
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NuCornea (Biosynthetic corneas) (Experimental): 6 patients will receive biosynthetic corneas when undergoing corneal transplantation
  Interventions: Device: NuCornea
- Donated human corneas (Active Comparator): 6 patients will receive a donated human cornea when undergoing corneal transplantation
  Interventions: Device: donated human corneas

INTERVENTIONS:
Device: NuCornea — Deep anterior lamellar corneal transplantation where the NuCornea is substituting a donor cornea
  Other Names: Biosynthetic cornea
  Arms: NuCornea (Biosynthetic corneas)
Device: donated human corneas — Deep anterior lamellar corneal transplantation with a donated cornea as graft material.
  Arms: Donated human corneas

SUMMARY:
Constructs made from cross-linked Human Recombinant Collagen type III are being used instead of human donor corneas in 6 patients at Deep anterior lamellar cornea grafting. Six patients serve as controls and are receiving human donor corneas using the same surgical technique. The twelve patients will be recruited from the local waiting list for patients to be undergoing corneal grafting. If the patients meet the inclusion criteria and agree to participate following oral and written consent, they will be randomized to either group. The patients will be followed for 12 months and documented with OCT, In Vivo Confocal Microscopy, slit lamp photography a o. The study is planned as a safety study with initial efficacy documentation.

DETAILED DESCRIPTION:
12 patients will be recruited from the waitinglist for corneal transplantation.The will all be of the age of 18 years or older and capable of making their own decisions. Their medical history and present medication is reveiwed and they undergo a thorough ophthalmological examination in order to find out if they meet the inclusion criteria and create baseline values for the study. Their general health or medication should not affect the cornea or ocular surface. The Eye should be healthy with the exception of the disease indication for corneal grafting. The corneal endothelium should be healthy. Any opacification in the eye to be grafted should not reach the Descemets membrane. Visual acuity in the fellow eye should be good. If these criteria are met the patient recieve oral and written information of the study. If they agree to participate they will be randomized to either recieve biosynthetic corneas ( 6 patients) or they will recieve a donated cornea ( 6 patients) . They will be scheduled for surgery within 2 weeks from the examination irrespective if they participate in the study or not.

The surgery will be anterior deep lamellar using the femtosecond laser to do the patient cut. The laser cut wil be done in topical anaaestesi. The remaining surgery with either be performed in local oor general anaestesia according to the patients wish. The diameter of the cut will be 7 mm in diameter. The graft material will be punched to a diameter of 7.25 mm. The thickness of the material will be 500 µm . An amniotic membrane will be placed on the top of the biosynthetic material and sutured with single stiches together with the graft.A bandage lens will be placed . The donated corneas will be sutured with singled about 8 stiches.

The biosynthetic corneas will recieve topical antibiotics and dexametasone for 8 weeks when the sutures, remnants of the amniotic membrane and the bandage lens is removed. The donated corneas will recieve topical dexametasone for 5 months and the sutures will be removed after 6 months.

The check-up Schedule will be at 1 day,1,2 weeks,1,,2 months and extra when needed.The protocol in these check-ups will be descriptive and the exyes will be documented with slit lamp photography. Epitelialisation will be monitored with fluorescein staining.

At the 3,6,9 and12 months will be extensive and the same in both groups. UCVA and BSCVA will be measured and also BCLCVA at 12 months. Corrneal topography,thickness sensitivity,tear production Visante OCT and slit- lamp photography will be performed. Tear samples will be taken also form earlier check-ups for proteomic analysis. In vivo confocal microscopy will be performed. The different examination with few exceptions can all be presented in results that can be quantified and statistically analysed.

The CRFs and the adverse report forms will be filled out both on computer forms and on paper.

The safety outcome criteria are: Good engraftment, maintained integrity of the graft, epithelialisation, transparency,no induced inflammation,no induced vasculatisation.

The preliminary efficacy criteria are: UCVA,BSCVA and BCLCVA

ELIGIBILITY:
Inclusion Criteria:

* Indication for Deep anterior lamellar corneal transplantation.
* No topical Eye medication.

Exclusion Criteria:

* No Eye disease other than the indication for the corneal graft.
* No general disease that might affect the cornea.
* No general medication that might affect the cornea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Biocompatibility: Good engraftment,epithelialization, no neovascularization,retained transparency, no host inflammatory reaction | 1 year
  Device replacing human donor cornea at Deep anterior lamellar transplantation.

SECONDARY OUTCOMES:
Visual acuity | 1 year
  Best spectacle corrected visual acuity,Best contactlens corrected Visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Per Fagerholm, MD,PhD, Principal Investigator — Dept of Ophthalmology, University Hospital, Linköping,Sweden